CLINICAL TRIAL: NCT00891241
Title: A Multi-Center, Single Dose, Phase I, Dosimetry, Biodistribution, and Safety Trial of LMI 1195-101 in Healthy Subjects and Patients With Heart Failure
Brief Title: A Phase 1 Trial to Determine Dosimetry, Biodistribution and Safety of LMI 1195-101 in Healthy Subjects and Patients With Heart Failure
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Lantheus Medical Imaging (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: LMI 1195 -101
Record Dates: First submitted 2009-04-29; First posted 2009-05-01 (Estimated); Last update posted 2020-11-16 (Actual); Status verified 2020-11

CONDITIONS: Heart Failure
Keywords: Heart Failure, PET Imaging, Implantable Cardioverter-Defibrillator, Dosimetry
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1 (Experimental): Healthy Population
  Interventions: Drug: LMI 1195-101
- Cohort 2 (Experimental): Heart Failure Subjects with a documented ejection fraction of 35% or less, and a diagnosis of NYHA Class II-III heart failure, history of ventricular arrhythmia and ICD placement
  Interventions: Drug: LMI 1195-101

INTERVENTIONS:
Drug: LMI 1195-101 — Single dose, bolus IV injection of LMI 1195
  Other Names: LMI 1195-101 Clinical Trial

SUMMARY:
The purpose of this clinical study is to estimate the safety and radiation dosimetry of a single dose of LMI1195 in healthy subjects and heart failure patients undergoing positron emission tomography (PET)

ELIGIBILITY:
Cohort 1 Inclusion:

* Healthy, age 18-40

Cohort 1 Exclusion:

* Significant or chronic medical illness
* Pregnant females
* Smoking within one month of enrollment
* Use of any prescription drugs within 4 weeks prior to dosing

Cohort 2 Inclusion:

* 30-70 year old subjects with a diagnosis of NYHA Class II-III heart failure
* Ejection fraction less than or equal to 35%
* Rest SPECT imaging within 90 days prior to enrollment

Cohort 2 Exclusion:

* Significant or chronic medical illness
* Pregnant females
* Known history of arrhythmogenic disorder or rhythm disorder

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-08; Primary Completion 2009-11 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Safety of LMI 1195 in terms of treatment-related adverse events | 14 days
  Number of study subjects exhibiting treatment-related adverse events

SECONDARY OUTCOMES:
Radiation Dosimetry of a single dose of LMI 1195 | 2 days
  Radiation dose to organs defined by the MIRD model, in mGy/MBq

CONTACTS AND LOCATIONS:
Overall Officials: L. Veronica Lee, M.D., Study Director — Medical Monitor - Lantheus Medical Imaging
Locations (2):
- United States (2):
  - Hartford Hospital, Hartford, Connecticut
  - Yale University Medical Center, New Haven, Connecticut